CLINICAL TRIAL: NCT00679341
Title: A Randomized, Multicenter, Phase ii Study of the Efficacy and Safety of Trastuzumab-MCC-DM1 vs. Trastuzumab (Herceptin®) and Docetaxel (Taxotere®) in Patients With Metastatic HER2-positive Breast Cancer Who Have Not Received Prior Chemotherapy for Metastatic Disease
Brief Title: A Study of the Efficacy and Safety of Trastuzumab Emtansine (Trastuzumab-MCC-DM1) vs. Trastuzumab (Herceptin®) and Docetaxel (Taxotere®) in Patients With Metastatic HER2-positive Breast Cancer Who Have Not Received Prior Chemotherapy for Metastatic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21976; TDM4450g (Other: Genentech)
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: HER2-positive breast cancer; HER2; Herceptin; Taxotere; MBC; Breast cancer; TDM1; TDM-1; HER2-positive; HER2+; HER2 positive breast cancer; HER2+ breast cancer; Armed Herceptin; Trastuzumab emtansine; Trastuzumab DM1
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Trastuzumab; Docetaxel

ARMS (2):
- Trastuzumab emtansine (Experimental): Patients received trastuzumab emtansine 3.6 mg/kg intravenously (IV) administered over 30-90 minutes every 3 weeks on Day 1 of each 21-day cycle.
  Interventions: Drug: Trastuzumab emtansine [Kadcyla]
- Trastuzumab + docetaxel (Active Comparator): Patients received a loading dose of trastuzumab 8 mg/kg IV + docetaxel 75 or 100 mg/m^2 IV on Day 1 of Cycle 1 followed by trastuzumab 6 mg/kg IV + docetaxel 75 or 100 mg/m^2 IV on Day 1 of all subsequent 21-day cycles.
  Interventions: Drug: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Trastuzumab emtansine [Kadcyla] — The total dose depended on the patient's weight on Day 1 of each cycle. Trastuzumab emtansine was administered every 3 weeks until investigator-assessed radiographic or clinical progressive disease (or until second disease progression for patients who crossed over), unacceptable toxicity, or study closure, whichever occurred first.
  Other Names: trastuzumab-DM1; trastuzumab-MCC-DM1; T-DM1
  Arms: Trastuzumab emtansine
Drug: Trastuzumab — The dose of trastuzumab was recalculated if body weight changed by more than ±10% from baseline. Trastuzumab was administered every 3 weeks until investigator-assessed radiographic or clinical progressive disease, or unmanageable toxicity. Patients in the trastuzumab + docetaxel arm who discontinued study treatment because of progressive disease were eligible to cross-over to trastuzumab emtansine treatment until a second progressive disease event, clinical deterioration, and/or intolerance.
  Other Names: Herceptin
  Arms: Trastuzumab + docetaxel
Drug: Docetaxel — Docetaxel was given at a dose of 75 or 100 mg/m^2 based on the investigator's decision. Patients in the trastuzumab + docetaxel arm who discontinued study treatment because of progressive disease were eligible to cross-over to trastuzumab emtansine treatment until a second progressive disease event, clinical deterioration, and/or intolerance.
  Other Names: Taxotere
  Arms: Trastuzumab + docetaxel

SUMMARY:
This was a Phase II, randomized, multicenter, international, 2-arm, open-label clinical trial designed to explore the efficacy and safety of trastuzumab emtansine (T-DM1) relative to the combination of trastuzumab and docetaxel in patients with human epidermal growth factor receptor 2 (HER2)-positive, unresectable, locally advanced breast cancer and/or metastatic breast cancer who have not received prior chemotherapy for metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with locally advanced or metastatic disease, and a candidate for chemotherapy.
* Human epidermal growth factor receptor 2 (HER2)-positive.
* No prior chemotherapy for their metastatic breast cancer (MBC).
* Measurable disease.
* Age ≥ 18 years.
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective, non-hormonal form of contraception or 2 effective forms of non-hormonal contraception by the patient and/or partner. Contraception use must continue for the duration of study treatment and for at least 6 months after the last dose of study treatment. Male patients whose partners are pregnant should use condoms for the duration of the study.

Exclusion Criteria:

* History of any chemotherapy for MBC.
* An interval of < 6 months from the completion of cytotoxic chemotherapy in the neo-adjuvant or adjuvant setting until the time of metastatic diagnosis.
* Trastuzumab ≤ 21 days prior to randomization.
* Hormone therapy < 7 days prior to randomization.
* Current peripheral neuropathy of Grade ≥ 3.
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those previously mentioned.
* Previous radiotherapy for the treatment of unresectable, locally advanced or metastatic breast cancer is not allowed if more than 25% of marrow-bearing bone has been irradiated or the last fraction of radiotherapy has been administered within approximately 3 weeks prior to randomization.
* Brain metastases that are untreated, symptomatic, or require therapy to control symptoms or any radiation, surgery, or other therapy to control symptoms from brain metastases within 2 months prior to randomization.
* History of exposure to the following cumulative doses of anthracyclines: Doxorubicin or liposomal doxorubicin > 500 mg/m^2; epirubicin > 900 mg/m^2; mitoxantrone > 120mg/m^2 and idarubicin > 90 mg/m^2.
* Current unstable angina.
* History of symptomatic congestive heart failure, or ventricular arrhythmia requiring treatment.
* History of myocardial infarction within 6 months prior to randomization.
* Left ventricular ejection fraction (LVEF) below 50% within approximately 28 days prior to randomization.
* History of decreased LVEF or symptomatic congestive heart failure (CHF) with previous adjuvant trastuzumab treatment.
* Cardiac troponin I ≥ 0.2 ng/mL within 28 days of randomization.
* Severe dyspnea at rest because of complications of advanced malignancy or requiring current continuous oxygen therapy.
* Current severe, uncontrolled systemic disease (eg, clinically significant cardiovascular, pulmonary, or metabolic disease; wound healing disorders; ulcers; or bone fractures).
* Major surgical procedure or significant traumatic injury within approximately 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment.
* Current pregnancy or lactation.
* History of receiving any investigational treatment within approximately 28 days prior to randomization.
* Current known infection with human immunodeficiency virus (HIV), active hepatitis B and/or hepatitis C virus.
* History of intolerance (including Grade 3-4 infusion reaction) or hypersensitivity to trastuzumab, murine proteins, or docetaxel.
* Known hypersensitivity to any of the study drugs, including the excipients, or any drugs formulated in polysorbate 80.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Guardino, MD/PhD, Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Perez EA, Hurvitz SA, Amler LC, Mundt KE, Ng V, Guardino E, Gianni L. Relationship between HER2 expression and efficacy with first-line trastuzumab emtansine compared with trastuzumab plus docetaxel in TDM4450g: a randomized phase II study of patients with previously untreated HER2-positive metastatic breast cancer. Breast Cancer Res. 2014 May 23;16(3):R50. doi: 10.1186/bcr3661. PMID 24887458
- [Derived] Hurvitz SA, Dirix L, Kocsis J, Bianchi GV, Lu J, Vinholes J, Guardino E, Song C, Tong B, Ng V, Chu YW, Perez EA. Phase II randomized study of trastuzumab emtansine versus trastuzumab plus docetaxel in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer. J Clin Oncol. 2013 Mar 20;31(9):1157-63. doi: 10.1200/JCO.2012.44.9694. Epub 2013 Feb 4. PMID 23382472

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel
Started | 67 | 70
Completed | 14 | 19
Not Completed | 53 | 51
Not completed — Disease progression | 42 | 36
Not completed — Adverse Event | 5 | 6
Not completed — Subject/guardian decision to discontinue | 3 | 0
Not completed — Death | 1 | 1
Not completed — Other | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Not treated | 0 | 2
Not completed — Physician/patient decision to withdraw | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel | Total
Number analyzed (Participants) | 67 | 70 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.6) | 52.1 (10.7) | 53.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 70 | 137
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) by the Investigator Using Modified Response Evaluation Criteria In Solid Tumors (RECIST)
Description: PFS was defined as the time from randomization (R) to first documented investigator-assessed radiographic or clinical disease progression (PD) or death due to any cause, whichever occurred first. For target lesions (TL), PD was defined as at least a 20% increase in the sum of the longest diameter (SLD) of TLs, taking as reference the SLD recorded since treatment started or the appearance of 1 or more new lesions. For non-TLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. Data for patients without PD or death were censored at the last date of tumor assessment prior to crossover (or, if no tumor assessment was performed after Baseline, at the R date +1 day). Data for patients who were lost to follow-up were censored at the last date of tumor assessment prior to crossover at which the patient was known to be progression free. Data for patients with no post-baseline tumor assessment were censored at the R date +1 day.
Time Frame: Baseline through the data cut-off date of 15 Nov 2010 (up to 2 years, 2 months)
Population: Intent-to-treat population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel
Number analyzed (Participants) | 67 | 70
Months | 14.2 [10.6 to NA] — The upper limit of the 95% confidence interval was not reached because of insufficient events. | 9.2 [8.2 to 11.2]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to the date of death from any cause. Patients who were alive at the time of analysis were censored at the date on which they were last known to be alive. Patients with no post-baseline were censored at the date of randomization plus 1 day.
Time Frame: Baseline through the data cut-off date of 31 Aug 2011 (up to 2 years, 11 months)
Population: Intent-to-treat population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel
Number analyzed (Participants) | 67 | 70
Months | NA [NA to NA] — The median and the upper and lower confidence intervals were not reached because of insufficient events. | NA [25.6 to NA] — The median and the upper confidence intervals were not reached because of insufficient events.

3. Secondary Outcome: Objective Response Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: A patient had an objective response if they had a complete response or a partial response on 2 consecutive occasions ≥ 4 weeks apart. For target lesions, a complete response was defined as the disappearance of all target lesions; a partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. For non-target lesions, a complete response was defined as the disappearance of all non-target lesions; a partial response was defined as the persistence of 1 or more non-target lesions.
Time Frame: Baseline through the data cut-off date of 15 Nov 2010 (up to 2 years, 2 months)
Population: All randomized patients with measureable disease at Baseline.
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel
Number analyzed (Participants) | 67 | 69
Percentage of patients | 64.2 [51.8 to 74.8] | 58.0 [45.5 to 69.2]

4. Secondary Outcome: Duration of Objective Response Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Duration of objective response was defined as the time from initial response to investigator-assessed radiographic or clinical disease progression or death on study from any cause. For target lesions, disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, disease progression was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Target lesions should be selected on the basis of their size (those with the longest diameter) and their suitability for accurate repeated measurements by imaging techniques or clinically. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions.
Time Frame: Baseline through the data cut-off date of 15 Nov 2010 (up to 2 years, 2 months)
Population: All randomized patients with measureable disease at Baseline. Only patients with an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel
Number analyzed (Participants) | 43 | 40
Months | NA [15.0 to NA] — The median and the upper confidence intervals were not reached because of insufficient events. | 9.5 [6.6 to 10.6]

5. Secondary Outcome: Clinical Benefit (CB) Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: CB was defined as an objective response (complete response [CR], partial response [PR]) or stable disease (SD) for 6 months after randomization. For target lesions (TL), CR=the disappearance of all TL; PR=at least a 30% decrease in the sum of the longest diameter (LD) of TL, taking as reference the baseline sum LD; SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started; PD=at least a 20% increase in the sum of the LD of TL, taking as reference the smallest sum of the LD recorded since the treatment started or the appearance of 1 or more new lesions. For non-TL, CR=the disappearance of all non-TL; PR=the persistence of 1 or more non-TL; SD=the persistence of 1 or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits; PD=the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TL.
Time Frame: Baseline through the data cut-off date of 15 Nov 2010 (up to 2 years, 2 months)
Population: All randomized patients with measurable disease at Baseline.
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel
Number analyzed (Participants) | 67 | 69
Percentage of patients | 74.6 [63.2 to 84.2] | 81.2 [70.7 to 89.1]

6. Secondary Outcome: Time to Symptom Progression
Description: Time to symptom progression was defined as the time from randomization to the first documentation of a ≥ 5-point decrease from baseline in the Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) subscale score of the Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire. The FACT-B questionnaire is a valid and reliable measure of symptoms associated with breast cancer. The TOI-PFB is a 24-item subscale generated using 3 subsections (Physical Well-Being [7 items], Functional Well-Being [7 items], and Additional Concerns [10 items]) from the FACT-B questionnaire. Patients responded to each item on a scale of 0-4 (Not at all-Very much). The total score ranged from 0 to 96. A higher score indicates fewer symptoms. A positive change score indicates improvement.
Time Frame: Baseline through the data cut-off date of 15 Nov 2010 (up to 2 years, 2 months)
Population: All randomized patients with a Baseline and at least 1 post-Baseline valid score.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel
Number analyzed (Participants) | 65 | 67
Months | 7.5 [4.2 to 15.1] | 3.5 [2.1 to 6.5]

7. Secondary Outcome: Serum Concentrations (Area Under the Concentration-time Curve [AUC]) of Trastuzumab Emtansine and Total Trastuzumab
Description: Serum samples were collected from all 67 patients enrolled in the trastuzumab emtansine arm using sparse pharmacokinetic sampling. Blood samples were collected prior to dosing and 30 minutes post-infusion of trastuzumab emtansine at Cycles 1 and 5. Serum samples were assayed for trastuzumab emtansine and total trastuzumab (sum of unconjugated trastuzumab and emtansine conjugated to trastuzumab) in indirect sandwich ELISAs. The area under the concentration-time curve (AUC) was estimated based on non-compartmental analysis using WinNonlin (Version 5.2.1) software.
Time Frame: Baseline through Cycle 5 (up to 4 months)
Population: Pharmacokinetic evaluable population: Patients who had adequate concentration-time data to estimate at least 1 pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: day•μg/mL
Groups:
- Trastuzumab Emtansine 3.6 mg/kg: Patients received trastuzumab emtansine 3.6 mg/kg intravenously (IV) administered over 30-90 minutes every 3 weeks on Day 1 of each 21-day cycle.
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 67
day•μg/mL
  Trastuzumab emtansine Cycle 1 (n=62) | 495 (158)
  Trastuzumab emtansine Cycle 5 (n=39) | 473 (141)
  Total trastuzumab Cycle 1 (n=60) | 700 (260)
  Total trastuzumab Cycle 5 (n=38) | 788 (323)

8. Secondary Outcome: Plasma Concentration of Free Emtansine
Description: Plasma samples were collected from all 67 patients in the trastuzumab emtansine group 30 minutes post-infusion of trastuzumab emtansine at Cycles 1 and 5. The plasma samples were assayed for free emtansine in a mass-spectrometric assay.
Time Frame: Baseline through Cycle 5 (up to 4 months)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Trastuzumab Emtansine 3.6 mg/kg
Number analyzed (Participants) | 67
ng/mL
  Cycle 1 (n=62) | 5.11 (2.34)
  Cycle 5 (n=39) | 4.71 (2.25)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization until 30 days following the last treatment, until the early termination visit, or until treatment-related adverse events resolved or stabilized, whichever occurred first.
Description: Safety population: All randomized patients who received at least 1 dose of study treatment. In the trastuzumab + docetaxel (T+D) group, 2 patients received no treatment and 2 patients received a dose of trastuzumab emtansine (TE) and were included in that group for safety analyses, resulting in 66 patients in the T+D group and 69 in the TE group.
Arm/Group | Trastuzumab Emtansine | Trastuzumab + Docetaxel
Serious Adverse Events (participants affected / at risk) | 14/69 | 17/66
Other Adverse Events (participants affected / at risk) | 66/69 | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=69) | Trastuzumab + Docetaxel (N=66)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 6
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 0
Cellulitis (Infections and infestations) | 0 | 2
Arthritis infective (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=69) | Trastuzumab + Docetaxel (N=66)
Neutropenia (Blood and lymphatic system disorders) | 11 | 43
Anaemia (Blood and lymphatic system disorders) | 9 | 18
Leukopenia (Blood and lymphatic system disorders) | 7 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 4
Palpitations (Cardiac disorders) | 4 | 2
Lacrimation increased (Eye disorders) | 5 | 13
Conjunctivitis (Eye disorders) | 5 | 3
Dry eye (Eye disorders) | 6 | 0
Nausea (Gastrointestinal disorders) | 34 | 29
Diarrhoea (Gastrointestinal disorders) | 11 | 30
Vomiting (Gastrointestinal disorders) | 17 | 17
Constipation (Gastrointestinal disorders) | 16 | 15
Stomatitis (Gastrointestinal disorders) | 8 | 13
Dyspepsia (Gastrointestinal disorders) | 11 | 8
Abdominal pain upper (Gastrointestinal disorders) | 12 | 4
Dry mouth (Gastrointestinal disorders) | 11 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Toothache (Gastrointestinal disorders) | 2 | 7
Gingival bleeding (Gastrointestinal disorders) | 4 | 0
Oral pain (Gastrointestinal disorders) | 0 | 4
Fatigue (General disorders) | 34 | 30
Pyrexia (General disorders) | 28 | 15
Oedema peripheral (General disorders) | 7 | 28
Asthenia (General disorders) | 16 | 14
Mucosal inflammation (General disorders) | 4 | 12
Chills (General disorders) | 10 | 5
Chest pain (General disorders) | 6 | 4
Pain (General disorders) | 2 | 5
Influenza like illness (General disorders) | 5 | 1
Nasopharyngitis (Infections and infestations) | 11 | 10
Upper respiratory tract infection (Infections and infestations) | 10 | 8
Urinary tract infection (Infections and infestations) | 5 | 11
Sinusitis (Infections and infestations) | 7 | 5
Influenza (Infections and infestations) | 5 | 2
Pharyngitis (Infections and infestations) | 4 | 3
Bronchitis (Infections and infestations) | 1 | 5
Rhinitis (Infections and infestations) | 5 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 4
Contusion (Injury, poisoning and procedural complications) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 30 | 4
Alanine aminotransferase increased (Investigations) | 18 | 4
Blood alkaline phosphatase increased (Investigations) | 10 | 2
Blood lactate dehydrogenase increased (Investigations) | 6 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 0
Platelet count decreased (Investigations) | 4 | 0
Weight increased (Investigations) | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 13 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Headache (Nervous system disorders) | 28 | 12
Dysgeusia (Nervous system disorders) | 6 | 15
Neuropathy peripheral (Nervous system disorders) | 10 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 14
Paraesthesia (Nervous system disorders) | 6 | 11
Dizziness (Nervous system disorders) | 3 | 6
Hypoaesthesia (Nervous system disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 8 | 12
Anxiety (Psychiatric disorders) | 6 | 5
Depression (Psychiatric disorders) | 5 | 4
Dysuria (Renal and urinary disorders) | 1 | 4
Breast pain (Reproductive system and breast disorders) | 1 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 44
Rash (Skin and subcutaneous tissue disorders) | 12 | 15
Nail disorder (Skin and subcutaneous tissue disorders) | 7 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 8
Erythema (Skin and subcutaneous tissue disorders) | 2 | 5
Acne (Skin and subcutaneous tissue disorders) | 6 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 4
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 4
Hypertension (Vascular disorders) | 9 | 6
Hot flush (Vascular disorders) | 0 | 10
Lymphoedema (Vascular disorders) | 3 | 5
Flushing (Vascular disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.